CLINICAL TRIAL: NCT05326919
Title: The Patient Cohort of the National Center for Precision Medicine in Leukemia
Acronym: eTHEMA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210850
Record Dates: First submitted 2022-01-28; First posted 2022-04-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; High-risk Myelodysplastic Syndrome; Secondary Myelofibrosis in Myeloproliferative Disease; Myeloproliferative Neoplasm, Unclassifiable
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute myeloid Leukemia (AML): Standard and routine care.
  For storage,limited volumes of blood or bone marrow aspirate will be added to usual sampling and stored.
  Interventions: Other: Biobanking
- Acute lymphoblastic leukemia (ALL): Standard and routine care.
  For storage,limited volumes of blood or bone marrow aspirate will be added to usual sampling and stored.
  Interventions: Other: Biobanking
- High-risk myelodysplastic syndrome (MDS): Standard and routine care.
  For storage,limited volumes of blood or bone marrow aspirate will be added to usual sampling and stored.
  Interventions: Other: Biobanking
- Myeloproliferative neoplasm -related myelofibrosis: Standard and routine care.
  For storage,limited volumes of blood or bone marrow aspirate will be added to usual sampling and stored.
  Interventions: Other: Biobanking

INTERVENTIONS:
Other: Biobanking — For storage,limited volumes of blood or bone marrow aspirate will be added to usual sampling and stored.

SUMMARY:
If for years the treatment strategy of leukemia and related disorders (LRDs, including acute leukemias and predisposition syndromes) has been based solely on whether the patient could receive or not intensive chemotherapy and transplantation, the advent of new targeted or less targeted drugs has led to the development of a growing number of new therapeutic approaches, very often offered to specific patient/disease subsets, justifying the generic term of 'precision medicine'.

As an international leukemia center of excellence, THEMA, the French National Center for Precision Medicine in Leukemia (selected as IHUB-2 by the French National Agency for Research), is a care, research, transfer and education initiative located at the Saint-Louis Research Institute (IRSL) in Paris and devoted to precision medicine in leukemia in a real-life environment.

The present non-interventional study (eTHEMA) is a pillar of the whole THEMA project. As a prerequisite for precision medicine, this program focuses on individual data collection, aiming to collect high-quality data not only in patients treated into prospective clinical trials, but in every THEMA patient with a special interest in outpatients' care and research.

The primary objective of this non-interventional study is to describe the baseline characteristics planned treatments and outcomes of patients newly diagnosed with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), high-risk myelodysplastic syndrome (MDS), or myeloproliferative neoplasm (MPN)-related myelofibrosis, when managed and treated according to standard diagnosis and care practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed previously untreated de novo, secondary or therapy-related leukemia or related disorders (LRD), including AML, ALL, HR-MDS (according to the international score IPSS), and MNP-related myelofibrosis
* Patient informed and not opposed to participating
* Affiliation to social security or any health insurance

Exclusion Criteria:

* LRD which is not morphologically proven (patients with granulocytic sarcoma may be included)
* Previous treatment for LRD, apart from:

  * Hydroxyurea or previous MDS/MPN-CML therapy in AML patients
  * Steroids, vincristine, intrathecal prophylactic or curative injection or previous CML therapy in ALL patients
  * Erythroid stimulating agents (ESAs), luspatercept, granulocyte colony-stimulating factor (G-CSF), eltrombopag or other TPO agonist, iron chelation therapy, hypomethylating agents (HMAs), lenalidomide or any investigational drug previously used to treat MDS in HR-MDS patients
  * Hydroxyurea, standard or pegylated interferon alpha, ruxolitinib or other JAK inhibitors, busulfan, anagrelide, ESAs or any investigational drug previously used to treat MPN in MPN-related myelofibrosis patients
* Patient under guardianship / curatorship
* Patient under AME
* Opposition of the patient to be enrolled in the eTHEMA cohort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), high-risk myelodysplastic syndrome (MDS), or myeloproliferative neoplasm (MPN)-related myelofibrosis, when managed and treated according to standard diagnosis and care practices
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2042-03 (Estimated); Study Completion 2042-03 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | at 5 years
Relapse Free Survival | at 5 years
Overall Survival | at 5 years

SECONDARY OUTCOMES:
Standardized evaluation of hematological response | After induction cycle which is between between day 25 and day 42 for patients treated intensively and between Month 1 and Month 6 for patients treated treated with low intensity regimen
Standardized evaluation of hematological response | After first consolidation cycle which is between 1 and 2 months
Standardized evaluation of hematological response | After last consolidation cycle which is between 3 and 8 months
Standardized evaluation of hematological response | Before HSCT
Standardized evaluation of hematological response | at day 100 after HSCT
Standardized evaluation of hematological response | at 5 years
Minimal measurable residual disease (MRD) response | After induction which is between day 25 and day 42 for patients treated intensively and between month 1 and month 6 for patients with low intensity regimen
Minimal measurable residual disease (MRD) response | After first consolidation cycle which is between 1 and 2 months
Minimal measurable residual disease (MRD) response | After last consolidation cycle which is between 3 and 8 months
Minimal measurable residual disease (MRD) response | Before HSCT
Minimal measurable residual disease (MRD) response | at day 100 after HSCT
Minimal measurable residual disease (MRD) response | at 5 years
Incidence of allogeneic HSCT | at 5 years
Modalities of allogeneic HSCT | at 5 years
Incidence of hematological relapses | at 5 years
Type of hematological relapses | at 5 years
Incidence of hematological progressions | at 5 years
Type of hematological progressions | at 5 years
Incidence of MRD relapses | at 5 years
Incidence of MRD progressions | at 5 years
Proportions of patients with treatment-related toxicities | at 5 years
  Treatment-related toxicities will be Evaluated by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Cumulative incidences of relapse | at 5 years
Cumulative incidences of non-relapse mortality | at 5 years
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at inclusion
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at the end of induction which is between day 25 and day 42 for patients treated intensively and between month 1 and month 6 for patients with low intensity regimen
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire.Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | after 2 consolidations courses which is between 3 months and 8 months
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire. Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at 3 months after the end of treatment
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire. Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at 6 months after the end of treatment
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire. Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at 12 months after the end of treatment
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire. Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality-of-life assessed using the EORTC-QLQ-C30 v3 questionnaire | at day 100 after hematopoietic stem cell transplant
  Quality-of-life will be assessed using the EORTC-QLQ-C30 v3 questionnaire. Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Incidence of secondary cancer | at 5 years
Incidence of secondary cancer | up to 15 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Avicenne, Bobigny
  - Hopital Robert Debré, Paris
  - Hôpital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao LP, Dumas-Rivero T, Barette L, Aguinaga L, Cheffai A, Chauvel C, Dal Bello R, Raffoux E, Clappier E, Duchmann M, Fenaux P, Lemaire P, Mathis S, Sebert M, Ades L, Itzykson R. Prognostic significance of monocytic-like phenotype in patients with AML treated with venetoclax and azacytidine. Blood Adv. 2025 Jul 22;9(14):3556-3565. doi: 10.1182/bloodadvances.2024015734. PMID 40249917